CLINICAL TRIAL: NCT02060448
Title: Exploring Two Emotion-Focused Treatment Modules in Non-Suicidal Self-Injury
Brief Title: Treatment Study for Non-Suicidal Self-Injury
Acronym: NSSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kate H. Bentley, Doctoral Candidate, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F31MH100761 (NIH); F31MH100761 (NIH)
Record Dates: First submitted 2014-02-07; First posted 2014-02-12 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Self Injurious Behavior Without Suicidal Intent
Keywords: Non-suicidal self-injury; Self-injurious behavior; NSSI; Anxiety; Depression; Transdiagnostic; CBT; Unified Protocol
MeSH Terms: conditions — Self-Injurious Behavior; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 2wk baseline + awareness (+ reappraisal) (Experimental): Participants in this arm will first undergo a two-week baseline phase. Participants who evidence a significant decrease in non-suicidal self-injurious thoughts and behaviors, or SITBs, (i.e., "responders") after emotion awareness training will go straight to a four-week follow-up, and not receive cognitive reappraisal. Participants who evidence a less than satisfactory response in non-suicidal SITBs (i.e., "partial responders") after emotion awareness training will return to a two-week baseline phase before receiving cognitive reappraisal, and then enter a four-week follow-up. Participants who evidence little to no response in non-suicidal SITBs (i.e., "non-responders") after emotion awareness training will immediately receive cognitive reappraisal and then enter a four-week follow-up.
  Interventions: Behavioral: Emotion awareness training; Behavioral: Cognitive reappraisal
- 2wk baseline + reappraisal (+ awareness) (Experimental): Participants will first undergo a two-week baseline phase. Participants who evidence a significant decrease in non-suicidal SITBs (i.e., "responders") after cognitive reappraisal will go straight to a four-week follow-up, and not receive emotion awareness training. Participants who evidence a less than satisfactory response in non-suicidal SITBs (i.e., "partial responders") after cognitive reappraisal will return to a two-week baseline phase before receiving emotion awareness training, and then enter a four-week follow-up. Participants who evidence little to no response in non-suicidal SITBs and behaviors (i.e., "non-responders") after cognitive reappraisal will immediately receive emotion awareness training and then enter a four-week follow-up.
  Interventions: Behavioral: Emotion awareness training; Behavioral: Cognitive reappraisal
- 4wk baseline + awareness (+ reappraisal) (Experimental): Participants in this arm will first undergo a four-week baseline phase. Participants who evidence a significant decrease in non-suicidal SITBs (i.e., "responders") after emotion awareness training will go straight to a four-week follow-up, and not receive cognitive reappraisal. Participants who evidence a less than satisfactory response in non-suicidal SITBs (i.e., "partial responders") after emotion awareness training will return to a two-week baseline phase before receiving cognitive reappraisal, and then enter a four-week follow-up. Participants who evidence little to no response in non-suicidal SITBs (i.e., "non-responders") after emotion awareness training will immediately receive cognitive reappraisal and then enter a four-week follow-up.
  Interventions: Behavioral: Emotion awareness training; Behavioral: Cognitive reappraisal
- 4wk baseline + reappraisal + (awareness) (Experimental): Participants in this arm will first undergo a four-week baseline phase. Participants who evidence a significant decrease in non-suicidal SITBs (i.e., "responders") after cognitive reappraisal will go straight to a four-week follow-up, and not receive emotion awareness training. Participants who evidence a less than satisfactory response in non-suicidal SITBs (i.e., "partial responders") after cognitive reappraisal will return to a two-week baseline phase before receiving emotion awareness training, and then enter a four-week follow-up. Participants who evidence little to no response in non-suicidal SITBs (i.e., "non-responders") after cognitive reappraisal will immediately receive emotion awareness training and then enter a four-week follow-up.
  Interventions: Behavioral: Emotion awareness training; Behavioral: Cognitive reappraisal

INTERVENTIONS:
Behavioral: Emotion awareness training — Four weekly individual treatment sessions focused on increasing awareness of one's emotions.
Behavioral: Cognitive reappraisal — Four weekly individual treatment sessions focused on thinking about stimuli in a way that diminishes one's emotions.

SUMMARY:
The overall aim of this study is to begin establishing an effective treatment for individuals who engage in non-suicidal self-injury (NSSI), as there are currently no evidence-based treatments that directly target this problematic behavior. Existing treatments that have demonstrated initial promise in reducing NSSI consist of many skills embedded in complex programs; therefore, the skill(s) responsible for improvements in NSSI are not clear. Procedures that focus on one's emotions, particularly that aim to increase emotional awareness and engagement in cognitive reappraisal (i.e., a way of thinking that lessens emotions), may be critical in effective NSSI treatment. The specific goals of this study are to investigate the effects of two specific emotion-focused treatment elements on NSSI. Participants will be ten individuals who meet the proposed Diagnostic and Statistical Manual for Mental Disorders, 5th edition (DSM-5; American Psychiatric Association) criteria for NSSI disorder and engage in NSSI to reduce or escape from negative emotions. Two core modules of the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders (UP; Barlow et al., 2011) will be adapted and delivered with the aim of reducing participants' non-suicidal self-injurious thoughts and behaviors. Each treatment module will consist of four 50-minute individual weekly sessions of emotion awareness training or cognitive reappraisal. The study will use a single-case experimental design, and phase change will be determined based on each participant's changes in non-suicidal self-injurious thoughts and behaviors.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Engage in non-suicidal self-injury (NSSI) to reduce or lessen negative thoughts or feelings
* Not taking psychotropic medications, or meet criteria for stability on a particular dose and are willing to maintain a stable dosage throughout the study
* Meet the proposed Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria for NSSI disorder, which includes:

  1. five or more days in which the individual has engaged in NSSI in the past year
  2. NSSI is associated with at least two two of the following: psychological precipitant (e.g., negative feelings or thoughts), urge prior to the act, preoccupation with NSSI, contingent response (e.g., expectation that the act will relieve a negative feeling state)
  3. clinically significant distress or interference caused by NSSI or its consequences
  4. NSSI does not occur exclusively during states of psychosis, delirium, or intoxication
  5. absence of suicidal intent

Exclusion Criteria:

* Current suicidal ideation and intent
* Currently receiving cognitive-behavioral therapy (CBT) or any psychotherapy to address NSSI, anxiety, depression, or other Axis I disorders (and are not willing to discontinue that treatment)
* Unwilling to refrain from initiating additional treatment during the course of the study
* Current or very recent symptoms that warrant immediate clinical attention, alternative treatment, and/or a higher level of care that cannot be provided through the study (e.g., florid delusions or hallucinations, rapid mood state, severe manic symptoms)
* Current or recent (within 3 months) history of substance use disorder (exception would be marijuana, caffeine, nicotine)
* Emotional symptomatology is due to a medical/physical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Frequency of non-suicidal self-injurious thoughts and behaviors | Daily (up to 126 days)
  Frequency of non-suicidal self-injurious thoughts and behaviors will be indicated by participants' responses to electronic questions delivered through a smart phone daily, assessed up to 126 days.

SECONDARY OUTCOMES:
Overall Anxiety Severity and Impairment Scale (OASIS) | Weekly (up to 18 weeks)
Overall Depression Severity and Impairment Scale (ODSIS) | Weekly (up to 18 weeks)
Beck Anxiety Inventory (BAI) | Weekly (up to 18 weeks)
Beck Depression Inventory (BDI-II) | Weekly (up to 18 weeks)
Deficits in Emotion Regulation Scale (DERS): Emotion Awareness and Nonacceptance of Negative Emotional Responses subscales | Weekly (up to 18 weeks)
Southampton Mindfulness Questionnaire (SMQ) | Weekly (up to 18 weeks)
Multi-dimensional Experiential Avoidance Questionnaire (MEAQ): Distraction/Suppression subscale | Weekly (up to 18 weeks)
Emotion Regulation Questionnaire (ERQ) | Weekly (up to 18 weeks)
Insomnia Severity Index (ISI) | Weekly (up to 18 weeks)
  Only three items of the ISI are included.
Subjective Symptoms Scale (SSS) | Weekly (up to 18 weeks)

OTHER OUTCOMES:
Self-Injury Implicit Association Test (SI-IAT) | up to 18 weeks
  The SI-IAT is a computerized behavioral test measures the implicit associations individuals hold about non-suicidal self-injury.

CONTACTS AND LOCATIONS:
Overall Officials: Kate H Bentley, M.A., Principal Investigator — Boston University; David H Barlow, Ph.D., Principal Investigator — Boston University
Locations (1):
- Center for Anxiety and Related Disorders, Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617